CLINICAL TRIAL: NCT03277443
Title: Accuracy of Computer Guided Surgery (vs) Conventional Model Surgery in Treatment of Skeletal Open Bite: A Randomized Clinical Trial
Brief Title: Accuracy of Computer Guided Surgery (vs) Conventional Model Surgery in Treatment of Skeletal Open Bite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ammar Ribhi Abu shama (Other)
Responsible Party: Sponsor-Investigator, Ammar Ribhi Abu shama, PHD Doctor in Oral and Maxillofacial Surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 292017
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Apertognathia
Keywords: Skeletal open bite
MeSH Terms: conditions — Open Bite | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: SM and VSM
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Model Surgery (Active Comparator): Lateral Cephalogram with analysis and tracing of facial profile.
  Modified model surgical tecnique:
  1. Obtain wax bite registration.
  2. Record face-bow transfer.
  3. Duplication of articulating model for surgical simulation.
  4. Measure all casts and bases in standard model surgery fashion.
  5. Fabricate intermediate splint & Final splint.
  6. Condylar repositional splint.
  Interventions: Procedure: Conventional model surgery; Device: 2D cephalometric radiograph
- Computer guided surgery (Experimental): Preoperative surgical simulation and immediate postoperative evaluation will be carried out using Multi Slice CT scan.
  Computer-aided planning for study group:
  All planning will be done using specialized software (Anatomage Invivo 5.3) for preoperative surgical simulation and immediate postoperative evaluation.
  Pre-operative Fabrication of computer aided surgical splint:
  In the study group a stereo splint will be fabricated using rapid prototyping (RP) technique to guide the osteotomy and another one will be fabricated after virtual osteotomy to guide the surgical cuts. And stent for guided holes.
  So that the osteotomy will be accomplished by the aid of computer guided templates that simulates the proper bite achieved preoperatively during surgical simulation and Planning.
  Interventions: Procedure: Computer guided surgery; Device: 3D computerized tomography

INTERVENTIONS:
Procedure: Computer guided surgery — Preoperative surgical simulation and immediate postoperative evaluation will be carried out using Multi Slice CT scan.Craniofacial images from 3D computerized tomography (3D-CT scan) can be used to create a 3D model, which can in turn be used for 3D Cephalometry measurements and surgical simulation.The process of 3D-model contains mounting of 3D virtual models in a 3D virtual articulator; and repositioning of 3D virtual models according to the STO then Fabrication of a 3D virtual intermediate surgical wafer; and materialization of the surgical wafer using a stereolithographic technique. The 3D model can produce actual movement of surgical cuts and movement of segments accordingly
  Arms: Computer guided surgery
Procedure: Conventional model surgery — preparation for orthognathic surgery which involves diagnosis with 2D cephalometric radiograph, face-bow transfer and model surgery on plaster dental cast, and fabrication of intermediate and final occlusal splint.
  Arms: Conventional Model Surgery
Device: 2D cephalometric radiograph — 2D cephalometric radiograph
  Arms: Conventional Model Surgery
Device: 3D computerized tomography — 3D computerized tomography
  Arms: Computer guided surgery

SUMMARY:
In patient with skeletal open bite, Dose computer-aided surgery enhances the clinical outcomes and accuracy versus conventional model surgery

DETAILED DESCRIPTION:
P Adult Patients with skeletal open bite.

I Computer guided surgery.

C Conventional articulating model surgery

O Outcome measure:

Outcome Name Measuring Device Measuring Unit (mm)

O1 Accuracy

Computer guided: Super-imposition of virtual surgery over the post- operative CT Scan composite models ( millimeter mm)

Conventional : Super-imposition of scanned articulator with mounted casts in the pre-planned mock surgery over post-operative scanned mounted occlusion ( millimeter mm)

O2 Anterior open Bite Closure

Standardized Multi Scan CT (millimeter mm)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from skeletal open bite caused by vertical posterior maxillary excess and/or short mandible ramus.
* Patients should be free from any systemic disease that may affect normal healing, and predictable outcome.
* Required two jaws orthographic surgery

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may retard the osteotomy healing.
* Patient with bad oral hygiene.
* Uncontrolled Diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-02-20 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of movement of surgical segments in millimeter | up to 4 months
  Computer guided Super-imposition of virtual surgery over the post- operative CT Scan composite models (millimeter mm).
  Conventional Super-imposition of scanned articulator with mounted casts in the pre-planned mock surgery over post-operative scanned mounted occlusion- accuracy would be compared by difference between Intervention and control in (millimeter mm).

SECONDARY OUTCOMES:
Anterior open Bite Closure (positive overbite in millimeter) | up to 4 months
  Standardized pre-surgery movement in amount of anterior open bite closure (mm) will be determined clinically and by radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa K Ezz, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided